CLINICAL TRIAL: NCT02266758
Title: Comparing Two Gestational Diabetes Screening Methods: A Pragmatic Outpatient RCT
Brief Title: Randomizing Two Gestational Diabetes Screening Methods in a Diverse HMO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kaiser Permanente (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: R01HD074794 (NIH); R01HD074794 (NIH)
Record Dates: First submitted 2014-05-22; First posted 2014-10-17 (Estimated); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Gestational Diabetes; Obesity; Pregnancy
Keywords: Gestational Diabetes; Obesity; Pregnancy
MeSH Terms: conditions — Diabetes, Gestational; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GDM Screening Method 1 (Other): GDM Screening Methods
  Interventions: Other: GDM Screening Methods
- GDM Screening Method 2 (Other): GDM Screening Methods
  Interventions: Other: GDM Screening Methods

INTERVENTIONS:
Other: GDM Screening Methods

SUMMARY:
This project randomizes two different screening strategies for diabetes in pregnancy, among a study population of over 17,500 pregnant women and their babies (over 35,000 total) in a large diverse health maintenance organization (HMO), to determine how diagnosis and treatment based on these two strategies in routine clinical care affects complications for the baby and the mother.

DETAILED DESCRIPTION:
Two recent randomized placebo-controlled trials show that gestational diabetes (GDM) treatment (vs. none) improves maternal and perinatal outcomes, based on diagnosis with a 2- step screening strategy. Also, a large multi-center prospective cohort study showed a linear relationship with glucose and maternal and perinatal outcomes, based on screening with a single 75g oral glucose tolerance test (OGTT). Based on this large cohort's findings, the American Diabetes Association recommended that clinical practice adopt the 1-step 75g screening approach for diagnosing GDM. The American College of Obstetrics & Gynecology took the opposite stance, recommending the traditional 2-step screening: because it alone has RCT outcome evidence. What is urgently needed to best inform clinical practice and health policy is not an additional GDM treatment vs. control trial, but a pragmatic randomized controlled trial (RCT) testing the 2 recommended clinical strategies. To pragmatically address this critical research gap, we propose to randomize an estimated 17,626 diverse women to GDM screening (2-step vs. 75g OGTT) as part of their clinical care in the Kaiser Permanente Northwest (KPNW) and Hawaii (KPH) regional health plans. The investigators will use the plans' electronic medical record (EMR) system at the time of GDM screening to randomize the women. Both KPNW and KPH regions universally screen for GDM at 24-28 weeks gestation, as part of clinical care. By randomizing GDM screening in the context of clinical care, the investigators will: Compare GDM prevalences (Aim 1) and differences in maternal and perinatal outcomes between screening strategies (Aim 2). Determine the concordance of the 75g OGTT with GDM diagnosed by 2-step, among a recruited sub-sample of 1,000 pregnant women at KPNW and KPH (Aim 3). The results of this pragmatic RCT are expected to help resolve the current public policy debate on the potential benefits and risks of each strategy in clinical obstetric practice.

ELIGIBILITY:
Inclusion Criteria:

* pregnant adult women in KPNW and KPH

Exclusion Criteria:

* pre-existing diabetes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23792 (Actual)
Dates: Start 2014-06-03 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Pregnancies with GDM diagnosis | During Pregnancy to Delivery, up to 10 months
  Diagnosis of GDM based on laboratory values for each screening approach (1-step or 2-step) as planned in the original protocol.
Number of Newborns with Large for Gestational Age (LGA) Birthweight | Birth
  Birthweight > 90th percentile
Number of neonates with any component of a composite perinatal outcome | Birth to first year of life
  Includes any of the following: number of neonatal deaths, stillbirths, shoulder dystocia, bone fracture, or nerve palsy
Number of pregnant women with Gestational Hypertension & Pre-Eclampsia | During Pregnancy to Delivery, up to 10 months
  Based on International Classification of Diseases (ICD-10) diagnoses
Number of Cesarean Section Deliveries | During Pregnancy to Delivery, up to 10 months
  Primary Cesarean Section

SECONDARY OUTCOMES:
Birthweight | Birth
  Will evaluate macrosomia, large for gestational age (LGA), small for gestational age (SGA) and average birthweight. LGA remains a primary outcome.
Number of Pregnant Women with GDM Requiring Treatment | During Pregnancy to Delivery, up to 10 months
  Maternal GDM requiring insulin or oral hypoglycemic treatment (class A2GDM)
Neonatal respiratory distress | Birth to first year of life
  Number of pregnancies for which newborn has a diagnosis of neonatal respiratory distress syndrome; planned in the original protocol.
Neonatal jaundice requiring treatment | Birth to first year of life
  Number of pregnancies for which newborn has a diagnosis of jaundice and received jaundice treatment; planned in the original protocol.
Neonatal hypoglycemia | Birth to first year of life
  Number of pregnancies for which newborn has a diagnosis of neonatal hypoglycemia; planned in the original protocol.
Number of stillbirths | During Pregnancy to Delivery
  Stillbirth is a secondary outcome; miscarriages were excluded
Number of Neonatal Deaths | First week of life
  Death of newborn under age 7 days
Number of Infants with Shoulder Dystocia | Birth to first year of life
  Diagnosed by ICD-10
Number of Infant Bone Fractures or Nerve Palsies associated with delivery | Birth to first year of life
  Diagnosed by ICD-10

OTHER OUTCOMES:
Neonatal sepsis | Birth up to 1 year
  Safety outcome. Number of pregnancies for which newborn has a diagnosis of neonatal sepsis
Neonatal intensive care unit (NICU) admission | Birth up to 1 year
  Safety outcome. Number of pregnancies for which newborn is admitted to the NICU
Preterm delivery (both <37 weeks and <32 weeks of gestation) | Birth up to 1 year
  Safety outcome. Number of pregnancies in which delivery took place before 37 weeks of gestation; separately, number or pregnancies in which delivery took place before 32 weeks of gestation
Induction of labor | During Pregnancy to Delivery, up to 10 months
  Safety outcome. Number of pregnancies in which labor was induced
Gestational Weight Gain | Pre-pregnancy, 1st trimester, 2nd trimester, 3rd trimester and overall to delivery, up to 10 months
  Weight Gain During Pregnancy
Changes in pre-pregnancy to post-partum maternal weight | pre-pregnancy up to 1 year post-partum
  Maternal height and weight measurements to evaluate average weight retention post-partum compared to pre-pregnancy
Number of Pregnancies with Multiple Maternal and Child GDM-Associated Outcomes | Beginning of Pregnancy up to 10 years post-partum
  This pragmatic GDM screening RCT evaluates rates of multiple maternal and child GDM-associated outcomes with two standard-of-care screening strategies in a large population of pregnant women at two diverse HMO sites with routine universal screening for GDM. This first primary outcome encompasses the overarching goals of our pragmatic RCT, and other specific primary outcomes will be listed as subsequent primary outcome measures. This outcome was initially registered as an overall primary outcome and was intended (as stated in the study protocol) to include the number of pregnancies diagnosed with GDM based on laboratory values of the two screening approaches; the primary GDM diagnosis has been updated separately as a primary outcome as per protocol.
Number and Intensity of Utilization of Health Care Services | During Pregnancy to Delivery, up to 10 months
  Quantification of health care visits, labs, procedures, and pharmacy for each pregnant woman
Changes in childhood height and weight measures | Annually after birth up to 10 years
  We will evaluate childhood growth percentiles and trajectories, as well as incidence of childhood overweight and obesity
Number of mothers with post-partum diabetes | Annually after birth up to 10 years
  Development of post-partum diabetes by ICD-10 diagnoses and lab measurement
Number of women with Post-partum depression | Birth up to 1 year
  Based on maternal ICD-10 diagnoses and questionnaire assessment
Number of children with metabolic syndrome | Annually from birth up to 10 years
  Based on ICD-10 diagnoses and also measured components including blood pressure, lipid measurements, body mass index, and diabetes
Number of Vaginal Assisted Deliveries | Delivery
  vaginal deliveries requiring assistance, including forceps and vacuum extraction
Number of pregnant women with anxiety or depression | During Pregnancy to Delivery, up to 10 months
  Based on ICD-10 diagnoses and questionnaire assessment

CONTACTS AND LOCATIONS:
Overall Officials: Teresa A Hillier, MD, MS, Principal Investigator — KP Center for Health Resarch, NW & Hawaii

REFERENCES:
- [Derived] Hillier TA, Pedula KL, Ogasawara KK, Vesco KK, Oshiro CES, Lubarsky SL, Van Marter J. Further implications from a pragmatic randomized clinical trial of gestational diabetes screening: per-protocol and as-treated estimates. Am J Obstet Gynecol. 2021 Nov;225(5):581-583. doi: 10.1016/j.ajog.2021.08.006. Epub 2021 Aug 9. PMID 34384772
- [Derived] Hillier TA, Pedula KL, Ogasawara KK, Vesco KK, Oshiro CES, Lubarsky SL, Van Marter J. A Pragmatic, Randomized Clinical Trial of Gestational Diabetes Screening. N Engl J Med. 2021 Mar 11;384(10):895-904. doi: 10.1056/NEJMoa2026028. PMID 33704936